CLINICAL TRIAL: NCT00630994
Title: Phase II Trial of Low Dose Decitabine (Dacogen) in Patients With Primary Myelofibrosis and Post ET/PV Myelofibrosis
Brief Title: Low-Dose Decitabine in Treating Patients With Symptomatic Myelofibrosis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Stopped due to slow accrual
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000588839; P30CA015083 (NIH); MC0788 (Other: Mayo Clinic Cancer Center); NCI-2009-01330 (Registry Identifier: NCI-CTRO); 07-005296 (Other: Mayo Clinic IRB)
Record Dates: First submitted 2008-03-06; First posted 2008-03-07 (Estimated); Results first posted 2012-04-02 (Estimated); Last update posted 2015-12-30 (Estimated); Status verified 2012-11

CONDITIONS: Chronic Myeloproliferative Disorders; Secondary Myelofibrosis
Keywords: primary myelofibrosis; secondary myelofibrosis; essential thrombocythemia; polycythemia vera
MeSH Terms: conditions — Myeloproliferative Disorders; Primary Myelofibrosis; Thrombocythemia, Essential; Polycythemia Vera | interventions — Decitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Dacogen

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as decitabine, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing.

PURPOSE: This phase II trial is studying the side effects and how well low-dose decitabine works in treating patients with symptomatic myelofibrosis.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the efficacy and safety of low-dose decitabine in patients with symptomatic primary myelofibrosis (PMF) or post essential thrombocythemic (ET) or polycythemic vera (PV) myelofibrosis.
* Analyze the ability of this drug to decrease pathologic angiogenesis and other stromal reactive features intrinsic to PMF or post ET/PV myelofibrosis.

OUTLINE: Patients receive low-dose decitabine IV over 1 hour on days 1-5. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. Patients achieving partial remission, complete remission, or clinical improvement may receive up to 12 courses of decitabine in the absence of disease progression or unacceptable toxicity.

After completion of study therapy, patients are followed periodically for up to 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histological confirmation of primary myelofibrosis or post essential thrombocythemic or polycythemic vera myelofibrosis

  * Reticulin fibrosis ≥ grade 1
* Evaluable and symptomatic disease worthy of treatment, characterized by ≥ 1 of the following:

  * Anemia, defined as hemoglobin < 11 g/dL or erythrocyte transfusion dependence
  * Palpable and symptomatic splenomegaly (palpable and symptomatic hepatomegaly is acceptable if previously splenectomized)
  * Severe, disease-related constitutional symptoms, including ≥ 1 of the following:

    * Severe night sweats
    * Fevers
    * Weight loss
    * Bone pain
* Absence of t(9;22) by fluorescent in situ hybridization (FISH) or standard cytogenetics OR prior demonstration of a lack of this translocation

PATIENT CHARACTERISTICS:

* Eastern Co-operative Oncology Group (ECOG) performance status 0-3
* Absolute neutrophil count (ANC) ≥ 1,000/mm³
* Platelet count ≥ 50,000/mm³
* Creatinine ≤ 2.0 mg/dL
* Direct or total bilirubin ≤ 2.0 mg/dL
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3 times upper limit of normal (ULN) (≤ 5 times ULN if elevation is attributed to hepatic extramedullary hematopoiesis)
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Not incarcerated in a municipality, county, state, or federal prison
* No serious medical condition or psychiatric illness that would preclude signing the informed consent
* No condition that, in the opinion of the treating physician, places the patient at unacceptable risk for study participation or confounds the ability to interpret study data
* Able to adhere to the study visit schedule and other study requirements

PRIOR CONCURRENT THERAPY:

* No other concurrent chemotherapy (e.g., hydroxyurea, thalidomide, interferon alpha, anagrelide, or other myelosuppressive agent) or experimental therapy

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2008-03; Primary Completion 2009-08 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ruben A. Mesa, MD, Study Chair — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Four (4) patient was recruited from March 2008 to May 2009 at Mayo Clinic. This trial was permanently closed in September 2009 due to slow accrual.
Groups:
- Decitabine: 20 mg/m^2/day intravenous over one hour on days 1-5 out of 28 days of treatment cycle
Period: Overall Study
Arm/Group | Decitabine
Started | 4
Completed | 0
Not Completed | 4
Not completed — Adverse Event | 1
Not completed — Disease Progression | 1
Not completed — Lack of Efficacy | 1
Not completed — Other | 1

BASELINE CHARACTERISTICS:
Arm/Group | Decitabine
Number analyzed (Participants) | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.8 (6.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 3
Region of Enrollment [Number; unit: participants]
  United States | 4
Prior disease specific therapy (including drugs, stem cell transplant, or splenectomy) [Number; unit: participants]
  Yes | 2
  No | 2
Prior bleeding events felt to be related to underlying disease [Number; unit: participants]
  Yes | 0
  No | 4
Prior thrombosis [Number; unit: participants]
  Yes | 2
  No | 2
Category of Primary myelofibrosis [Number; unit: participants]
  Primary Myelofibrosis | 2
  Post Essential Thrombocythemia (ET) Myelofibrosis | 1
  Post Polycythemia Vera (PV) Myelofibrosis | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Achieve a Confirmed Response (Complete Remission (CR), Partial Remission (PR), or Clinical Improvement (CI)), According to International Working Group (IWG) Consensus Criteria.
Description: Confirmed response: objective status of CR, PR, or CI on 2 consecutive evaluations >=4 weeks apart.
  CR:Complete resolution of disease-related symptoms and signs; peripheral blood count remission; normal leukocyte differential; bone marrow histologic remission.
  PR: All criteria for CR except the bone marrow histologic remission. CI: one of the following in the absence of both disease progression and CR/PR: minimum (MI) 20-g/L increase (INC) in hemoglobin level; MI 50% reduction in palpable splenomegaly (>=10cm); MI 100% INC in platelet count(>=50000x10^9/L) or ANC (>=0.5x10^9/L)
Time Frame: Every 4 weeks during treatment (up to 16 weeks)
Population: All participants who met the eligibility criteria that have signed a consent form and went on treatment were evaluable for response. The study was terminated early due to slow enrollment. The primary outcome measure should be assessed with caution.
Measure: Number; unit: participants
Arm/Group | Decitabine
Number analyzed (Participants) | 4
participants | 1

2. Secondary Outcome: Overall Survival(OS)
Description: OS was defined as the time from registration to death of any cause.
Time Frame: up to 3 years
Population: Study terminated prematurely. Analysis not performed.
Arm/Group | Decitabine
Number analyzed (Participants) | 0

3. Secondary Outcome: Time to Disease Progression
Description: Time to disease progression is defined as the time from registration to progression of disease or death due to any cause.
  Progression was defined as any one or more of the following:
  1)progressive splenomegaly; 2) leukemic transformation confirmed by a bone marrow blast count of >= 20%; 3) an increase in peripheral blood blast percentage of >=20% that lasts for >= 8 weeks.
Time Frame: up to 3 years
Population: Study terminated prematurely. Analysis not performed.
Arm/Group | Decitabine
Number analyzed (Participants) | 0

4. Secondary Outcome: Number of Participants With Constitutional Symptoms
Description: Constitutional symptoms including the presence of one or more of the following felt to be attributed to the disease: severe night sweats, fevers, weight loss and bone pain. Symptoms were assessed every cycle during treatment.
Time Frame: Up to 48 weeks
Population: Study terminated prematurely. Analysis not performed.
Arm/Group | Decitabine
Number analyzed (Participants) | 0

5. Secondary Outcome: Number of Participants With Severe Adverse Events
Description: Severe adverse events were defined as grade 3 or higher, regardless of attribution to study drugs. Adverse events were graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 3. Adverse events were assessed every cycle during treatment.
Time Frame: Up to 48 weeks
Measure: Number; unit: participants
Arm/Group | Decitabine
Number analyzed (Participants) | 4
participants
  Anemia | 3
  Platelet count decreased | 1
  Neutrophil count decreased | 2
  Leukopenia | 1
  Alkaline Phosphatase Increased | 1
  Ascites | 1
  Clostridial Infection | 1
  Hyperglycemia | 1

ADVERSE EVENTS:
Arm/Group | Decitabine
Serious Adverse Events (participants affected / at risk) | 1/4
Other Adverse Events (participants affected / at risk) | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Decitabine (N=4)
Ascites (Gastrointestinal disorders) | 1 (1)
Clostridial infection (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Decitabine (N=4)
Anemia (Blood and lymphatic system disorders) | 4 (17)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (4)
Fatigue (General disorders) | 4 (16)
Alkaline phosphatase increased (Investigations) | 1 (1)
Bilirubin (Investigations) | 1 (1)
Leukopenia (Investigations) | 2 (5)
Neutrophil count decreased (Investigations) | 3 (7)
Platelet count decreased (Investigations) | 4 (12)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (3)

LIMITATIONS AND CAVEATS:
Study terminated early. Most analyses were not performed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes